CLINICAL TRIAL: NCT02584361
Title: Vestibular Function Evaluated by the Video Head Impulse Test (vHIT) and Vertigo Perceived by the Patients Before and After Cochlear Implant Surgery.
Brief Title: Cochlear Implant and Vestibular Function.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Leise Elisabeth Hviid Korsager, BSc, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47190
Record Dates: First submitted 2015-08-31; First posted 2015-10-22 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Sensorineural Hearing Loss; Deafness; Hearing Loss
Keywords: Hearing loss; Cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cochleostomy (Active Comparator): In this group the insertion of the electrode into cochlea will be performed by drilling a hole in cochlea (cochleostomy).
  Interventions: Procedure: Cochleostomy
- Round window approach (Active Comparator): In this group the insertion of the electrode into cochlea will be performed through an incision in the membrane (paracentesis) of the round window (round window approach = RWA)
  Interventions: Procedure: Round window approach

INTERVENTIONS:
Procedure: Round window approach — In this group the insertion of the electrode into cochlea will be performed through an incision in the membrane (paracentesis) of the round window (round window approach = RWA).
  Other Names: RWA
  Arms: Round window approach
Procedure: Cochleostomy — In this group the insertion of the electrode into cochlea will be performed by drilling a hole in cochlea (cochleostomy).
  Arms: Cochleostomy

SUMMARY:
This study investigate weather one type of cochlear implant (CI) surgery (insertion of the electrode via paracentesis of the round window (RWA)) leads to less vertigo than another type of CI surgery (cochleostomy). The participants will be randomized into 2 groups: RWA or cochleostomy. They will be examined with a video head impulse test (vHIT) before and after CI surgery to clarify their vestibular function.

DETAILED DESCRIPTION:
Cochlear implant is an advanced type of hearing advice. It consists of an outer microphone, which picks up sound and sends it through an electrode into the cochlear.

With a cochlear implant people, that are profoundly deaf or have severe hearing loss, can get their hearing back.

Vertigo is one of the most common side effects to cochlear implant surgery. In this study we will investigate if one type of CI surgery (insertion of the electrode via paracentesis of the round window) leads to less vertigo than another type of CI surgery (cochleostomy).

In the randomization there will be stratified according to age (60+/-), residual hearing (yes/no) and gain before surgery (+/-0,68). Three different surgeons will do the surgeries. All technical aspect of the surgery, other than the insertion of the electrode into cochlea, is being done identically.

Electrodes from Cochlear, MEDEL and AB is being used. We will compare the findings from the vHIT examination with the subject dizziness perceived of the patient.

The patients will be examined before surgery, the day after their surgery and one month after their surgery. The same examinator will perform all the vHIT tests. The test will be performed in continuation of the patient's other visits at the Department of Audiology and Department of Otorhinolaryngology -Head and Neck Surgery.

ELIGIBILITY:
Inclusion Criteria:

* deaf or severe hard of hearing
* normal or slightly affected vestibular function (gain >0,50)

Exclusion Criteria:

* subjects with otosclerosis
* subject who will have the CI surgery for preservation of the residual hearing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Vestibular function | 1 month
  Measured by video head impulse test one month after CI surgery in connection with consultation for CI activation

SECONDARY OUTCOMES:
Subjective dizziness | 1 month
  Measured by Dizziness Handicap Inventory Score (DHI).
Dizziness | 1 day
  Measured by a visuel analog scale (VAS) the day after cochlear implant surgery.
Dizziness | 1 month
  Measured by a visuel analog scale (VAS) in connection with consultation for CI activation.
T level | 1 month
  T level is a electropsysiological value. It is the minimum electrical signal in the electrode required for the patient to sense sound.
C level | 1 month
  C level is the maximum electrical signal in the electrode that is acceptable for the patient to tolerate the sound.
NRT level | 1 month
  Neural response telemetry, is an electrical response of the auditory nerve, when stimulated electrically.

CONTACTS AND LOCATIONS:
Overall Officials: Leise Korsager, BSc, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, DK-Odense, Denmark

REFERENCES:
- [Background] Wanscher JH, Faber CE, Grontved AM. [Cochlear implantation in deaf adults: effect on quality of life]. Ugeskr Laeger. 2006 Aug 14;168(33):2656-9. Danish. PMID 16942684
- [Background] Ovesen T, Johansen LV. Post-operative problems and complications in 313 consecutive cochlear implantations. J Laryngol Otol. 2009 May;123(5):492-6. doi: 10.1017/S0022215108003691. Epub 2008 Oct 10. PMID 18845035
- [Background] Todt I, Basta D, Ernst A. Does the surgical approach in cochlear implantation influence the occurrence of postoperative vertigo? Otolaryngol Head Neck Surg. 2008 Jan;138(1):8-12. doi: 10.1016/j.otohns.2007.09.003. PMID 18164986
- [Background] Krause E, Louza JP, Hempel JM, Wechtenbruch J, Rader T, Gurkov R. Effect of cochlear implantation on horizontal semicircular canal function. Eur Arch Otorhinolaryngol. 2009 Jun;266(6):811-7. doi: 10.1007/s00405-008-0815-5. Epub 2008 Sep 20. PMID 18807058
- [Background] Richard C, Fayad JN, Doherty J, Linthicum FH Jr. Round window versus cochleostomy technique in cochlear implantation: histologic findings. Otol Neurotol. 2012 Sep;33(7):1181-7. doi: 10.1097/MAO.0b013e318263d56d. PMID 22892806
- [Background] Sun CH, Hsu CJ, Chen PR, Wu HP. Residual hearing preservation after cochlear implantation via round window or cochleostomy approach. Laryngoscope. 2015 Jul;125(7):1715-9. doi: 10.1002/lary.25122. Epub 2015 Jan 13. PMID 25583631
- [Background] Macdougall HG, McGarvie LA, Halmagyi GM, Curthoys IS, Weber KP. The video Head Impulse Test (vHIT) detects vertical semicircular canal dysfunction. PLoS One. 2013 Apr 22;8(4):e61488. doi: 10.1371/journal.pone.0061488. Print 2013. PMID 23630593
- [Background] Havenith S, Lammers MJ, Tange RA, Trabalzini F, della Volpe A, van der Heijden GJ, Grolman W. Hearing preservation surgery: cochleostomy or round window approach? A systematic review. Otol Neurotol. 2013 Jun;34(4):667-74. doi: 10.1097/MAO.0b013e318288643e. PMID 23640087
- [Background] Zawawi F, Alobaid F, Leroux T, Zeitouni AG. Patients reported outcome post-cochlear implantation: how severe is their dizziness? J Otolaryngol Head Neck Surg. 2014 Dec 10;43(1):49. doi: 10.1186/s40463-014-0049-z. eCollection 2014. PMID 25492268